CLINICAL TRIAL: NCT03910192
Title: Mindfulness-based Coaching to Reduce Abnormal Nocturnal Hypertension in Atrial Fibrillation
Brief Title: Mindfulness to Reduce Ambulatory Hypertension in Atrial Fibrillation
Acronym: AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: York University (Other)
Collaborators: Southlake Regional Health Centre (Other)
Responsible Party: Principal Investigator, Paul Ritvo, Full Professor, York University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0031-1617
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Atrial Fibrillation; Hypertension; Mindfulness; Cardiovascular Risk Reduction
MeSH Terms: conditions — Atrial Fibrillation; Hypertension

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness meditation coaching (Experimental): Mindfulness-based coaching - participants will receive instructions on (a) mindfulness meditation and gentle mindful movement through home-based and in-class participation at the Southlake Cardiovascular Rehabilitation Clinic and (b) personal coaching support. The health coach will further assist participants through either face-to-face or telephone-based discussions. They will meet with the health coach at mutually-agreed upon on times for designated time periods.
  Interventions: Behavioral: Mindfulness-based coaching
- dietary cardiovascular risk reduction coaching (Active Comparator): Cardiovascular risk reduction education - No change to standard of care where participants will receive instructions (in person or by phone call) on how to integrate exercise and dietary changes in your lifestyle to reduce your risk of future cardiovascular events. These instructions will be centered around the DASH dietary practices.
  Interventions: Behavioral: Dietary cardiovascular risk reduction coaching

INTERVENTIONS:
Behavioral: Mindfulness-based coaching — 16 week mindfulness-based protocol focused on home-based and weekly group practice of mindfulness meditation and mindful movement.
  Arms: Mindfulness meditation coaching
Behavioral: Dietary cardiovascular risk reduction coaching — Regular in-person meetings, phone calls, or email from study coordinator instructing them on how to integrate exercise and dietary changes in their lifestyle to reduce their risk of future cardiovascular events.
  Arms: dietary cardiovascular risk reduction coaching

SUMMARY:
The aim of this study is to evaluate the effectiveness of a 16 week mindfulness-based coaching program compared to a cardiovascular risk reduction education program.

Both groups will undergo 24-hour ambulatory blood pressure monitoring, along with assessments of psychological measures (see bellow) at study baseline, midpoint (8 weeks), and conclusion (16 weeks).

In addition, both groups will also undergo 24-hour Holter monitoring assessments at study beginning and conclusion to assess possible episodes of atrial tachyarrhythmia during the assessed interval.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-80
* Diagnosed Atrial Fibrillation
* Night time (Sleep Time) Systolic Blood Pressure≥120 OR Daytime (awake) Systolic Blood Pressure ≥ 135
* Able and Willing to sign Informed Consent Form

Exclusion Criteria:

* Scheduled for Surgery

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-03-14 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Night time (Sleep) Systolic Blood Pressure | 16 weeks
  The primary outcome of this study will be change in ANBP from baseline when compared to subsequent follow-up study time points.
Daytime time (Awake) Systolic Blood Pressure | 16 Weeks
  The primary outcome of this study will be change in daytime ABP from baseline when compared to subsequent follow-up study time points.

SECONDARY OUTCOMES:
Nocturnal Dipping | 16 Weeks
  ANBP will be calculated as the percentage of nocturnal drop in systolic blood pressure in relation to its daytime values
Atrial Tachyarrhythmia Episodes | 16 Weeks
  24-hour Holter monitoring assessments using the MARS® ambulatory ECG system at baseline and 4 months to assess atrial tachyarrhythmia episodes lasting 30 seconds or more
Hospital Anxiety and Depression Scale (HADS) | 16 Weeks
  14 item self-report questionnaire evaluating anxiety and depression symptoms in medical populations
Profile of Mood States (POMS-SF) | 16 Weeks
  65 item self-report questionnaire examining mood and changes in mood over a period, POMS, in both original and shorter 37 item format, has been extensively used in clinical settings
Five Facet Mindfulness Questionnaire - Short Form (FFMQ-SF) | 16 Weeks
  24 item the magnitude and changes over time in mindfulness levels, including its five - observing, describing experience, acting with awareness, non-judging of inner experience, and nonreactivity to inner experience facets.
SF-12 v2 Health Survey | 16 Weeks
  assesses self reported physical and mental health, providing separate scores for 8 sub-domains of physical and mental health (e.g. physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health).
Pittsburgh Sleep Quality Index (PSQI) | 16 Weeks
  The instrument, widely used in epidemiological or clinical contexts, is comprised of seven sub-components (i.e. sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbance, medication use, and daytime dysfunction) leading to a global sleep quality score.
Cardiac Anxiety Questionnaire (CAQ) | 16 Weeks
  18 item index of HFA, a measure of anxiety sensitivity specific to cardiovascular patients. The CAQ conceptualizes HFA as a 3 dimensional measure, including heart-related fear, avoidance, attention subscales.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Ritvo, Ph.D, Principal Investigator — York Univrsity
Locations (1):
- Southlake Regional Health Centre, Newmarket, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No